CLINICAL TRIAL: NCT06908746
Title: Efficacy and Safety of Citrate Anticoagulation in CRRT for Patients With Liver Failure/DysfuncTION, the CAUTION Trial! A Retrospective Study on Etiology of Liver Failure and Their Complications
Acronym: Caution
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: Project ID 6806; Edge 003873 (Other: Antwerp University Hospital)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Liver Failure; AKI - Acute Kidney Injury
Keywords: CRRT; liver failure; AKI
MeSH Terms: conditions — Liver Failure; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study design A retrospective cohort study will be conducted to compare the efficacy and safety of citrate anticoagulation in CRRT among patients with liver failure/dysfunction and severe shock.

Objectives

1. Primary Objective: To determine if the etiology of liver failure impacts the incidence of citrate-related complications in patients undergoing CRRT.
2. Secondary Objectives: To compare the efficacy of citrate anticoagulation in terms of renal recovery, filter lifespan, and patient survival between those with liver failure/dysfunction and severe shock.

DETAILED DESCRIPTION:
Continuous renal replacement therapy (CRRT) is a crucial intervention for managing acute kidney injury (AKI) in critically ill patients. Citrate anticoagulation has become a preferred method in CRRT due to its effect in longer filter longevity and less bleeding compared to unfractionated heparin1. However, its use in specific patient populations, such as those with liver failure or severe shock, necessitates careful evaluation.

Citrate acts as an anticoagulant by chelating calcium, an essential cofactor in the coagulation cascade, thus preventing clot formation within the extracorporeal circuit2. The citrate-calcium complex is then metabolized mainly in the liver, where citrate is converted into bicarbonate, and calcium is released back into the bloodstream. This mechanism provides dual benefits: effective anticoagulation and metabolic alkalization.

Patients with liver failure present unique challenges for citrate anticoagulation. Impaired liver function can lead to the accumulation of citrate, resulting in high anion gap metabolic acidosis and hypocalcemia3. These risks underscore the need for vigilant monitoring and potential adjustment of citrate dosing in this population. The aim of the present study is to explore whether the etiology of liver failure, which can range from alcoholic liver disease to drug-induced liver injury or shock liver, influences the incidence and severity of citrate-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients diagnosed with AKI requiring CRRT. Caution Protocol V1.0 24-07-2024
* Documented liver failure or significant liver dysfunction (e.g., elevated liver enzymes, bilirubin levels, or clinical diagnosis of liver failure) and clincal diagnosis of shock (NE of 0.25 μg/kg/min and or association of second vasopressor).
* Age ≥ 18 years.

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients diagnosed with AKI requiring CRRT
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint: | During admission at ICU
  Incidence of citrate-related metabolic complications (e.g., citrate accumulation).

SECONDARY OUTCOMES:
Secondary Safety Endpoints | During admission at ICU
  * Incidence of electrolyte imbalances (e.g., hypocalcemia).
  * Incidence of adverse events related to anticoagulation.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jacobs, Dr., Principal Investigator — Antwerp Univesity Hospital
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs R, Verbrugghe W, Dams K, Roelant E, Couttenye MM, Devroey D, Jorens P. Regional Citrate Anticoagulation in Continuous Renal Replacement Therapy: Is Metabolic Fear the Enemy of Logic? A Systematic Review and Meta-Analysis of Randomised Controlled Trials. Life (Basel). 2023 May 17;13(5):1198. doi: 10.3390/life13051198. PMID 37240843
- [Background] Mehta RL, McDonald BR, Aguilar MM, Ward DM. Regional citrate anticoagulation for continuous arteriovenous hemodialysis in critically ill patients. Kidney Int. 1990 Nov;38(5):976-81. doi: 10.1038/ki.1990.300. No abstract available. PMID 2266683
- [Background] Kramer L, Bauer E, Joukhadar C, Strobl W, Gendo A, Madl C, Gangl A. Citrate pharmacokinetics and metabolism in cirrhotic and noncirrhotic critically ill patients. Crit Care Med. 2003 Oct;31(10):2450-5. doi: 10.1097/01.CCM.0000084871.76568.E6. PMID 14530750

DOCUMENTS (1):
  • Study Protocol (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/46/NCT06908746/Prot_000.pdf